CLINICAL TRIAL: NCT06937502
Title: The Relationship Between Functionality and Pain, Range of Motion, Neck Disability, and Quality of Life in Temporomandibular Disorders: A Cross-Sectional Study
Brief Title: Functionality and Clinical Correlates in TMD
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Elif Kabasakal, LECTURER, Istinye University
Other Study IDs: ISU-2025-003
Record Dates: First submitted 2025-04-20; First posted 2025-04-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Disorders (TMD); Functional Limitation; Pain Severity; Neck Disability; Quality of Life
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temporomandibular Disorders - Functionality Study Group: Mandibular functionality will be assessed using the Mandibular Function Impairment Questionnaire. Active temporomandibular joint (TMJ) range of motion (ROM) will be measured with a caliper. Pain will be evaluated using the Visual Analog Scale (VAS), neck disability using the Neck Disability Index (NDI), and quality of life using the World Health Organization Quality of Life Questionnaire (WHOQOL).

SUMMARY:
Temporomandibular disorders (TMD) are among the most common causes of orofacial pain and refer to structural and functional impairments related to the masticatory muscles, surrounding soft tissues, and/or the temporomandibular joint (TMJ). They negatively affect individuals physically, psychologically, and socially. The structural and functional impairments observed in TMD typically manifest as pain, restricted jaw movement, joint sounds, and muscle tension. In addition to these core symptoms, secondary issues such as chewing difficulties may also occur. Pain in TMD can negatively impact many orofacial functions, especially chewing. Functional impairment in individuals with TMD may result from pain, restricted jaw mobility, muscle tension, alterations in muscle activation, mandibular asymmetry, and morphological changes in the joint. These findings highlight the importance of addressing factors associated with functional impairment in individuals with TMD.

Pain severity is strongly associated with functional limitations of the TMJ and neck disability. Particularly in cases of muscular-origin TMD, significant impairments in neck muscle function and joint mobility have been observed. This condition directly affects jaw function and leads to a decrease in quality of life. The impact of TMD on quality of life is directly related to pain severity and functional limitations. As pain severity increases, limitations in daily activities and reductions in overall quality of life also increase. Therefore, a multidisciplinary approach to TMD is essential for pain management, functional rehabilitation, and improving quality of life.

The aim of this study is to investigate the relationships between functionality and pain, range of motion, neck disability, and quality of life in individuals with TMD. Understanding these relationships will form a basis for the effective management of TMD and improving individuals' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Aged between 18 and 55 years
* Diagnosed with temporomandibular disorders (TMD) and exhibiting at least one of the three main symptoms (jaw pain, limited mouth opening, and/or temporomandibular joint sound)
* A Mini-Mental State Examination (MMSE) score of 24 or higher
* Pain score of 3 or above on the Visual Analog Scale (VAS)

Exclusion Criteria:

* History of complex surgery, trauma, chemoradiotherapy, and/or tumors involving the head and neck region
* Ongoing use of analgesics, anti-inflammatory or psychiatric medications, and/or substance abuse
* Significant tooth loss that interferes with chewing function
* Use of dental prosthesis
* Ongoing tooth pain
* Receiving any TMD-specific treatment prior to or during the evaluation period
* History of orthodontic treatment
* Diagnosis of disc displacement without reduction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include individuals aged 18-55 diagnosed with temporomandibular disorders (TMD) who present at least one main symptom (jaw pain, limited mouth opening, or TMJ sounds), have a VAS pain score ≥3, and an MMSE score ≥24. Participation will be voluntary with informed consent.
  Exclusion criteria include history of head/neck surgery, trauma, cancer treatment, significant tooth loss, dental prosthesis use, ongoing tooth pain, current medication affecting pain perception, previous orthodontic or TMD-specific treatment, and diagnosis of disc displacement without reduction.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Temporomandibular Joint Functionality Assessment | At baseline
  The Mandibular Function Impairment Questionnaire (MFIQ) will be used to assess mandibular functionality. The MFIQ is designed to evaluate the patient's perception of mandibular functional impairment. It consists of 17 items, each rated on a 5-point Likert scale, with a total score ranging from 0 to 68. The questionnaire reflects the difficulty experienced during specific movements or tasks. Higher scores indicate greater functional impairment of the mandible.
Temporomandibular Joint Range of Motion Assessment | At baseline
  Active range of motion (ROM) will be evaluated. A caliper will be used to measure maximal mouth opening. For this assessment, the participant will be instructed to open their mouth as wide as possible. The movement will be repeated three times, and during the third repetition, the distance between the upper and lower central incisors will be measured and recorded.
Pain Assessment | At baseline
  The Visual Analog Scale (VAS) will be used to measure the intensity of pain. This scale includes numbers ranging from 0 to 10, where "0" indicates no pain and "10" represents the worst pain imaginable. The participant will be informed that the pain intensity increases along the scale from 0 to 10 and will be asked to mark the point that best represents the severity of pain they are experiencing.
Neck Disability Assessment | At baseline
  The Neck Disability Index (NDI) will be used to determine the level of neck disability in participants. The scale consists of ten items, covering topics such as neck pain intensity, personal care, lifting, reading, headaches, concentration, driving, sleeping, and recreational activities. Each item contains six response options that assess the degree of pain and limitation. Scoring ranges from 0 to 5 for each item, with a total score ranging from 0 to 50. Based on the total score, disability levels are classified as follows:
  0-4 = no disability, 5-14 = mild disability, 15-24 = moderate disability, 25-34 = severe disability, 35 and above = complete disability.
Quality of Life Assessment | At baseline
  The World Health Organization Quality of Life Scale (WHOQOL-BREF) evaluates five main domains: general health, physical health, psychological well-being, social relationships, and environment. It includes parameters such as pain, sleep, energy (physical health); positive feelings, self-esteem, body image (psychological health); social support and personal relationships (social health); and financial resources, transportation, safety, and access to healthcare (environmental health). The scale uses a 5-point Likert system, ranging from "1 = Very Dissatisfied" to "5 = Very Satisfied." Higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istınye University, Istanbul,, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided